CLINICAL TRIAL: NCT05599100
Title: Virtual Training for Latino Caregivers to Manage Symptoms of Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kaiser Permanente (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Magaly Ramirez, Assistant Professor, School of Public Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00013410; 5U54AG063546-04 (NIH)
Record Dates: First submitted 2022-10-23; First posted 2022-10-31 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-07

CONDITIONS: Caregiver Burden; Alzheimer Disease; Dementia; Behavioral Symptoms
MeSH Terms: conditions — Caregiver Burden; Alzheimer Disease; Dementia; Behavioral Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STAR-VTF (Experimental): Participants will receive the STAR-VTF intervention.
  Interventions: Behavioral: STAR-Caregivers Virtual Training & Follow-up (STAR-VTF)

INTERVENTIONS:
Behavioral: STAR-Caregivers Virtual Training & Follow-up (STAR-VTF) — For 6-8 weeks, caregivers will complete online training modules asynchronously. Caregivers will be instructed to complete one module per week. The content of the modules is as follows: Module 1 introduces caregivers to the behavioral treatment of dementia, realistic expectations, and effective communication; Module 2 covers the ABC (antecedents, behaviors, consequences) approach to problem-solving, including rationale and development of an ABC plan; Module 3 instructs caregivers to review the ABC plan and revise as needed; Module 4 covers pleasant events and managing negative thinking; Module 5 instructs caregivers to review the ABC plan, pleasant activities schedule, and to revise as needed; Module 6 covers coping with caregiving and maintaining gains. Each module takes about 45 minutes to complete. The modules use text, pictures, and illustrations with a voiceover presentation. Caregivers will receive the online training modules in their preferred language (English or Spanish).

SUMMARY:
The goal of this pilot study is to improve the STAR-Caregivers Virtual Training & Follow-up (STAR-VTF) intervention for Latino caregivers of people living with dementia. The main objectives are to: (1) culturally adapt STAR-VTF online training modules, (2) pilot test Latino caregivers' responses to the adapted online training modules, and (3) develop an online survey to collect caregiver outcomes in a future study. Participants will receive the STAR-VTF intervention and asked to complete online surveys and participate in an exit interview to provide feedback on their experience.

DETAILED DESCRIPTION:
The objectives of this study are to: (1) culturally and linguistically adapt the STAR-Caregivers Virtual Training & Follow-up (STAR-VTF) online training modules for Latino caregivers of people living with dementia (PLWD), (2) pilot test Latino caregivers' responses to the adapted online training modules, and (3) develop a REDCap survey to pragmatically collect caregiver outcomes in a future study.

The study will use a single-arm pilot trial design with Latino caregivers of PLWD. The investigators will assess self-reported outcomes at baseline and 6-8 weeks post-enrollment using a REDCap survey. Outcome measures will include the Revised Memory and Problem Behavior Checklist and Preparedness for Caregiving Scale. In addition, the investigators will assess caregivers' perceived usability of the online training modules and will conduct qualitative interviews 6-8 weeks post-enrollment. The interviews will assess caregiver satisfaction with and acceptability of the adapted online training modules.

The investigators expect to enroll up to 20 participants. The primary objective of this study is to pilot test the adapted online training modules. Therefore, it is not powered to detect an effect of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Lives with a person living with dementia (PLWD) or within 5 miles
* Provides at least 8 hours of care per week
* Self-identifies as Hispanic/Latino
* Caregiver self-report of PLWD having ≥ 3 behavioral and/or psychological symptoms of dementia occurring ≥ 3 in past week

Exclusion Criterion:

* PLWD lives in assisted living or skilled nursing facilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magaly Ramirez, PhD, MS, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Teri L, Truax P, Logsdon R, Uomoto J, Zarit S, Vitaliano PP. Assessment of behavioral problems in dementia: the revised memory and behavior problems checklist. Psychol Aging. 1992 Dec;7(4):622-31. doi: 10.1037//0882-7974.7.4.622. PMID 1466831
- [Background] Salvia MG, Dawidowski A, Schapira M, Figar S, Soderlund ME, Seinhart D, Camera L, Teri L. Spanish Revised Memory and Behavior Problems Checklist Scale (SpRMBPC): trans-cultural adaptation and validation of the RMBPC questionnaire. Int Psychogeriatr. 2011 Sep;23(7):1160-6. doi: 10.1017/S1041610210002073. Epub 2011 Feb 4. PMID 21294937
- [Background] Gutierrez-Baena B, Romero-Grimaldi C. Development and psychometric testing of the Spanish version of the Caregiver Preparedness Scale. Nurs Open. 2021 May;8(3):1183-1193. doi: 10.1002/nop2.732. Epub 2020 Dec 19. PMID 33340272
- [Background] Sevilla-Gonzalez MDR, Moreno Loaeza L, Lazaro-Carrera LS, Bourguet Ramirez B, Vazquez Rodriguez A, Peralta-Pedrero ML, Almeda-Valdes P. Spanish Version of the System Usability Scale for the Assessment of Electronic Tools: Development and Validation. JMIR Hum Factors. 2020 Dec 16;7(4):e21161. doi: 10.2196/21161. PMID 33325828

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | STAR-VTF
Started | 16
Completed | 15
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | STAR-VTF
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Preparedness for Caregiving Scale [Mean (Standard Deviation); unit: units on a scale] — Population: 2 participants were excluded from the analysis (1 was lost to follow up and the other did not respond to follow up outcome assessment)
  units on a scale
    number analyzed (Participants) | 14
    (all) | 1.98 (0.33)
Revised Memory and Behavior Problem Checklist (Overall Caregiver Reaction) [Mean (Standard Deviation); unit: units on a scale] — Population: 2 participants were excluded from the analysis (1 was lost to follow up and the other did not respond to follow up outcome assessment)
  units on a scale
    number analyzed (Participants) | 14
    (all) | 40.40 (16.48)

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline Revised Memory and Behavior Problem Checklist Score at 6 Weeks (Overall Caregiver Reaction)
Description: The Revised Memory and Behavior Problem Checklist is a 24-item scale measuring caregiver reaction to memory, depression, and disruptive behavior problems. Each item asks about a problem the care recipient is experiencing. For each problem the care recipient experiences, caregivers are asked to rate how much the problem upsets the caregiver on a Likert scale ranging from 0 (not at all) to 4 (extremely). Scores for caregiver reaction are calculated by taking the sum of the individual items. Total scores can range from 0 to 96, with higher scores reflect caregivers being more upset when memory and behavior problems happen.
  We report the change in scores by subtracting the total score at baseline from the total score at 6 weeks. The possible range for the change in total scores is from -96 to 96. A negative change indicates that caregivers' reaction has improved, while a positive change indicates that caregivers' reaction has worsened.
Time Frame: Change from baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STAR-VTF
Number analyzed (Participants) | 14
units on a scale | -6.90 (14.35)

2. Primary Outcome: Change in Baseline Preparedness for Caregiving Scale Score at 6 Weeks
Description: In the Preparedness for Caregiving Scale, caregivers rate how prepared they are for various aspects of caregiving. The instrument contains 8 items that ask caregivers how well prepared they believe they are to provide physical care, emotional support, deal with the stress of caregiving, and set up in-home support services. Each item is rated on a 5-point scale ranging from 0 (not at all prepared) to 4 (very well prepared). The score is calculated by taking the average of all items answered.
  We report the change in average scores by subtracting the average score at baseline from the average score at 6 weeks. The possible range for the change in average scores is from -4 to 4. A negative change indicates that caregivers' preparedness has worsened, while a positive change indicates that caregivers' preparedness has improved.
Time Frame: Change from baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | STAR-VTF
Number analyzed (Participants) | 14
score on a scale | 0.63 (0.73)

3. Secondary Outcome: System Usability Scale
Description: The System Usability Scale (SUS) is a 10-item questionnaire designed to assess the usability of and caregivers' satisfaction with the modules. Caregivers rate their agreement with statements on a 5-point scale, from "strongly disagree" to "strongly agree." A single score is calculated by converting each item's score to a 0-4 scale, summing the adjusted scores, and then multiplying by 2.5 to obtain a final score ranging from 0 to 100. Higher scores indicate better usability and caregiver satisfaction. General interpretive ranges suggest excellent usability (score of 85 and above), good usability (scores of 70-84), average usability (scores of 50-69), and poor usability (scores below 50).
Time Frame: Week 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STAR-VTF
Number analyzed (Participants) | 13
units on a scale | 77.8 (10.8)

4. Secondary Outcome: System Usability Scale
Description: as for outcome 3
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STAR-VTF
Number analyzed (Participants) | 12
units on a scale | 77.7 (12.9)

5. Secondary Outcome: System Usability Scale
Description: as for outcome 3
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STAR-VTF
Number analyzed (Participants) | 10
units on a scale | 74.6 (19.2)

6. Secondary Outcome: System Usability Scale
Description: as for outcome 3
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STAR-VTF
Number analyzed (Participants) | 13
units on a scale | 73.7 (16.3)

7. Secondary Outcome: System Usability Scale
Description: as for outcome 3
Time Frame: Week 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STAR-VTF
Number analyzed (Participants) | 12
units on a scale | 75.8 (14.3)

8. Secondary Outcome: System Usability Scale
Description: as for outcome 3
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STAR-VTF
Number analyzed (Participants) | 11
units on a scale | 79.2 (14.5)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | STAR-VTF
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT05599100/Prot_SAP_ICF_000.pdf